CLINICAL TRIAL: NCT02437487
Title: ECOSPOR: A RandomizEd, Double Blind, Placebo COntrolled, Parallel Group Study of SER 109 to Prevent Recurrent ClOstRidium Difficile Infection
Brief Title: SER-109 Versus Placebo to Prevent Recurrent Clostridium Difficile Infection (RCDI)
Acronym: ECOSPOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SERES-004
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Clostridium Difficile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SER-109 (Experimental): SER 109 (1 × 108 SporQs)
  Interventions: Drug: SER-109
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER-109 — SER 109 is a rationally designed ecology of bacterial spores enriched from stool donations obtained from healthy, screened donors.
  Other Names: Purified Eubacterial Spores, Encapsulated
  Arms: SER-109
Drug: Placebo — Placebo will be identical to the investigator product but will not contain product spores or non-spore solids. Placebo will consist of 92% glycerol and 8% normal saline.
  Arms: Placebo

SUMMARY:
The study will involve administering the study drug as a single dose of study drug or placebo. This study is designed to demonstrate the superiority of the experimental drug versus placebo in adult patients with recurrent CDI.

DETAILED DESCRIPTION:
ECOSPOR is a Phase 2, multicenter, randomized, double blind, placebo controlled clinical study with 2 treatment arms (SER-109 or placebo). Patients who have diarrhea and a positive C. difficile test result on a stool sample, and who have responded to standard of care antibiotic treatment will receive study drug on Day 1.

Those patients who experience a recurrence of CDI up to 8 weeks after SER 109 or placebo treatment will be offered an opportunity to enroll in an open label SER 109 extension study (Study SERES 005).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, indicating that the patient understands the purpose of and procedures required for the study. Patients who are unable to provide informed consent will not be included in the study.
2. Male or female patients ≥ 18 years.
3. ≥ 3 episodes of CDI within the previous 9 months, inclusive of the current episode with documentation of ≥ 2 episodes.

Exclusion Criteria:

1. Female patients who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.
2. Known or suspected toxic megacolon and/or known small bowel ileus.
3. Active irritable bowel syndrome with diarrhea within the previous 12 months.
4. Major gastrointestinal surgery (eg, significant bowel resection or diversion) within 3 months before enrollment (this does not include appendectomy or cholecystectomy) or any history of total colectomy or bariatric surgery.
5. History of inflammatory bowel disease (ulcerative colitis, Crohn's disease, microscopic colitis) with diarrhea believed to be caused by active inflammatory bowel disease in the past 24 months.
6. Admitted to or expected to be admitted to an acute care facility or intensive care unit for medical reasons (not just boarding). Patients discharged from an acute care facility before Day 1 or residing in nursing homes or rehabilitation facilities may be enrolled.
7. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (patients on maintenance chemotherapy may only be enrolled after consultation with medical monitor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Trucksis, Phd, MD, Study Director — Seres Therapeutics
Locations (30):
- United States (30):
  - North County Gastroenterology, Oceanside, California
  - University Of California Davis, Sacramento, California
  - Ventura Clinical Trials, Ventura, California
  - ZASA Clinical Research, Atlantis, Florida
  - Omega Research Consultants LLC, DeBary, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Emory University, Atlanta, Georgia
  - Idaho Falls Infection Diseases, Idaho Falls, Idaho
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Johns Hopkins Bayview Medical, Baltimore, Maryland
  - Metropolitan Gastroenterolgy Group Pc, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Cntr, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Chatfield, Minnesota
  - Sundance Clinical Research, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Englewood Hospital and Medical Center, Englewood Cliffs, New Jersey
  - Mount Sinai Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Regional Infectious Diseases-Infusion Center Inc, Lima, Ohio
  - Drexel University/Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Brown Alpert Medical School, Providence, Rhode Island
  - University of Texas School of Public Health, Houston, Texas
  - Medical Associates of Central Virginia, Lynchburg, Virginia

REFERENCES:
- [Derived] Bryant JA, Vulic M, Walsh EA, Allen EG Jr, Beauchemin NJ, Chafee ME, Diao L, Fenn K, Ford KA, Hasson BR, Litcofsky KD, Lombardo MJ, Martinez A, O'Brien EJ, Straub TJ, Sykes SM, Marshall LF, Winkler JA, McGovern BH, Ford CB, Wortman JR, Henn MR. The impact of an oral purified microbiome therapeutic on the gastrointestinal microbiome. Nat Med. 2026 Jan;32(1):186-196. doi: 10.1038/s41591-025-04076-w. Epub 2026 Jan 5. PMID 41491103
- [Derived] McGovern BH, Ford CB, Henn MR, Pardi DS, Khanna S, Hohmann EL, O'Brien EJ, Desjardins CA, Bernardo P, Wortman JR, Lombardo MJ, Litcofsky KD, Winkler JA, McChalicher CWJ, Li SS, Tomlinson AD, Nandakumar M, Cook DN, Pomerantz RJ, Aunins JG, Trucksis M. SER-109, an Investigational Microbiome Drug to Reduce Recurrence After Clostridioides difficile Infection: Lessons Learned From a Phase 2 Trial. Clin Infect Dis. 2021 Jun 15;72(12):2132-2140. doi: 10.1093/cid/ciaa387. PMID 32255488

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SER-109 | Placebo
Started | 59 | 30
Actual Treatment Received | 60 | 29
Intention-to-Treat Population | 59 | 30
Completed | 32 | 16
Not Completed | 27 | 14

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | SER-109 | Placebo | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 15 | 43
  >=65 years | 31 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (16.60) | 66.1 (14.02) | 64.5 (15.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 60
  Male | 19 | 10 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 54 | 29 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 27.72 (6.402) | 27.65 (5.744) | 27.70 (6.150)
Number of Previous CDI Episodes [Count of Participants; unit: Participants]
  1 | 0 | 0 | 0
  2 | 0 | 0 | 0
  3 | 28 | 20 | 48
  4 | 21 | 5 | 26
  5 or more | 10 | 5 | 15
Stool Frequency [Count of Participants; unit: Participants]
  0-2 per day | 0 | 0 | 0
  3 per day | 5 | 0 | 5
  4-5 per day | 27 | 12 | 39
  6-9 per day | 14 | 8 | 22
  10 or more per day | 11 | 8 | 19
  Unknown | 2 | 2 | 4
White Blood Cells Category [Count of Participants; unit: Participants]
  less than 12,000 | 18 | 7 | 25
  12,001 to 15,000 | 1 | 2 | 3
  15,001 or more | 0 | 0 | 0
  Unknown | 40 | 21 | 61
Albumin < 2.5 mg/dL [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 20 | 8 | 28
  Unknown | 38 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With CDI Recurrence
Time Frame: 8 weeks after treatment.
Population: Intention-To-Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 59 | 30
participants | 26 | 16
Statistical Analysis 1: Comparison: SER-109 vs Placebo; Test type: Superiority; Relative Risk = 1.2217, 95% CI 2-sided [0.7919 to 1.8849]

2. Secondary Outcome: Time to Recurrence of CDI
Description: Kaplan-Meier estimate of median number of days to recurrence
Time Frame: Recurrence of CDI up to 24 weeks after treatment.
Population: Intention to Treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 59 | 30
days | NA [35.0 to NA] — Insufficient number of participants with events. | NA [14.0 to NA] — Insufficient number of participants with events.

3. Secondary Outcome: Number of Subjects With CDI Recurrence
Time Frame: 4 Weeks
Population: Intention-to-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 59 | 30
Participants | 22 | 14
Statistical Analysis 1: Comparison: SER-109 vs Placebo; Test type: Superiority; Relative Risk = 1.2624, 95% CI 2-sided [0.7668 to 2.0785]

4. Secondary Outcome: Number of Subjects With CDI Recurrence
Time Frame: 12 Weeks
Population: Intention-to-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 59 | 30
Participants | 26 | 16
Statistical Analysis 1: Comparison: SER-109 vs Placebo; Test type: Superiority; Relative Risk = 1.2217, 95% CI 2-sided [0.7919 to 1.8849]

5. Secondary Outcome: Number of Subjects With CDI Recurrence
Time Frame: 24 Weeks
Population: Intention-to-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | SER-109 | Placebo
Number analyzed (Participants) | 59 | 30
Participants | 31 | 17
Statistical Analysis 1: Comparison: SER-109 vs Placebo; Test type: Superiority; Relative Risk = 1.0878, 95% CI 2-sided [0.7383 to 1.6029]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | SER-109 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/29
Serious Adverse Events (participants affected / at risk) | 9/60 | 3/29
Other Adverse Events (participants affected / at risk) | 33/60 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER-109 (N=60) | Placebo (N=29)
Drug Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basilic Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Worsening Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mental Status Changes due to Dehydration (Psychiatric disorders) | 1 (1) | 0 (0) — Secondary to Clostridium difficile infection
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) — Secondary to Clostridium difficile infection
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Acute On Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis of Left Lower Leg (Infections and infestations) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
CHF Exacerbation (Cardiac disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Worsening of Headache (Nervous system disorders) | 1 (1) | 0 (0)
LLE DVT (Vascular disorders) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute on Chronic Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Foot Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Cough (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Blockage of Dialysis Stunt (General disorders) | 1 (1) | 0 (0)
Enlarged Pelvic Mass (General disorders) | 1 (1) | 0 (0)
DVT Left Leg (Vascular disorders) | 1 (1) | 0 (0)
Metastatic Non Small Cell Lung Cancer (NSCLC) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Episode of Unresponsiveness (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Worsening of Generalized Weakness (General disorders) | 0 (0) | 1 (1) — Secondary to Clostridium difficile infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SER-109 (N=60) | Placebo (N=29)
Diarrhea (Gastrointestinal disorders) | 15 | 4
Abdominal Pain (Gastrointestinal disorders) | 13 | 4
Flatulence (Gastrointestinal disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications must be submitted to Sponsor for review at least 30 days prior to publication. Sponsor can require removal of confidential information other than study data and Site/Investigator agree to consider Sponsor's suggestions with respect to the presentation of study data. Sponsor can force publication to be deferred for a period of up to 60 days in order to file any patents.